CLINICAL TRIAL: NCT03735082
Title: The Efficacy and Safety of Apatinib Combined With Paclitaxel and Carbopatin Intensive Regimen in Neoadjuvant Therapy for Locally Advanced Triple-negative Breast Cancer :Single Arm, Phase II Clinical Trail
Brief Title: Apatinib Combined With Paclitaxel and Carbopatin Intensive Regimen in Neoadjuvant Therapy for Locally Advanced Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ004
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib+Paclitaxel+Carboplatin (Experimental): apatinib 250mg, d1-14,14day/cycle; Paclitaxel 175mg/m2,d1,14days/cycle; Carboplatin AUC=4,d1,14day/cycle
  Interventions: Drug: Apatinib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Apatinib — apatinib 250mg,qd,d1-14,14day/cycle
Drug: Paclitaxel — paclitaxel 175mg/m2,d1,14day/cycle+carboplatin AUC=4,d1,14day/cycle
Drug: Carboplatin — carboplatin AUC=4,d1,14day/cycle;

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Apatinib Combined With Paclitaxel and Carbopatin Intensive Regimen in Neoadjuvant Therapy for Locally Advanced Triple-negative Breast patients

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) has the characteristics of early onset, high malignancy, less treatment, and resistance to treatment. Advanced patients have shorter survival than other subtypes. Changes in traditional chemotherapy regimens for breast cancer (ie, the addition of carboplatin) are potential ways to improve patient outcomes. Although anthracyclines and cyclophosphamide play a very positive role in the treatment of breast cancer, there are also small and serious long-term risks. Anti-angiogenic drugs are currently one of the few targeted therapies that have achieved some efficacy in TNBC. Apatinib, a targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with breast cancer. Considering of current status of anti-angiogenic drugs in the field of breast cancer, results of apatinib in advanced breast cancer, and current unmet clinical needs, the investigator conducted this study to assess the efficacy and safety of Apatinib Combined With Paclitaxel and Carbopatin Intensive Regimen in Neoadjuvant Therapy for Locally Advanced Triple-negative Breast patients

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 year-old women;
2. Physical condition ECOG PS: 0-1;
3. Previously untreated, histologically or cytologically confirmed to be triple negative breast cancer;
4. Breast mass > 2cm, or ipsilateral lymph node metastasis (ipsilateral armpit, internal mammary, supraclavicle); Note: According to RECIST version 1.1, confirmed by CT or MRI,There must be at least one measurable lesion;If the target lesion is a lymph node requiring a short diameter greater than 1.5 cm, and the target lesion is not suitable for surgical treatment;
5. Laboratory tests meet the following criteria: absolute count of blood neutrophils (ANC) ≥1.5×109/L; platelet (PLT)≥100×109/L; hemoglobin (HB)≥10g/dl; serum bilirubin ≤ 1.5 times the upper limit of normal value; AKP,ALT and AST≤2.5 times the upper limit of normal value;AKP, ALT and AST≤5 times the upper limit of normal value when liver metastasis;Urea nitrogen ≤ 1.5 times the upper limit of normal value,serum creatinine ≤ 1.5 times the upper limit of normal value;
6. Expected survival time ≥ 3 months;
7. Women of child-bearing age should be carried out pregnancy test (serum or urine) within 7 days before recruit, the results should be negative; and are willing to adopt the appropriate methods of contraception during the trial;
8. Patients volunteered to join the study and signed informed consent.

Exclusion Criteria:

1. There are other metastasis sites other than ipsilateral lymph node metastasis (ipsilateral armpit, internal mammary, supraclavicular);
2. Have received anti-tumor treatment;
3. Patients with hypertension who are not well controlled by antihypertensive medication (systolic pressure >140 mmHg, diastolic pressure >90 mmHg); have uncontrolled or severe cardiovascular disease, such as Refractory angina pectoris,congestive heart failure occurred within 6 months prior to screening ; myocardial infarction occurred within 12 months before screening; any clinically significant ventricular arrhythmia history, prolonged QT interval; history of cerebrovascular accident, symptomatic and medication required Coronary heart disease;
4. Significant clinical dysfunction of the digestive tract may affect the intake, transport or absorption of oral medications (eg, inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
5. Patients with previous bleeding history, clinically significant bleeding symptoms, and patients with clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood + and above, vasculitis, etc.; urine protein positive patients;
6. Major surgery or severe traumatic injury, fracture, or poor healing wound within 4 weeks;
7. Allergic to apatinib and/or its adjuvants, paclitaxel, carboplatin, etc.;
8. Female patients during pregnancy or lactation, female patients with fertility and pregnancy test positive, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period
9. The patient has a severe concomitant disease, or any other condition the investigator believes is not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 3 months
  pCR defined as no invasive and non-invasive (DCIS) residuals in breast and armpit lymph nodes
safety of treatment: Incidence of adverse events | every 2 weeks
  Incidence of adverse events by maximum CTCAE grade (v4.03; NCI 2010)

SECONDARY OUTCOMES:
rate of breast-pCR | 3 months
  breast-pCR defined as no invasive and non-invasive (DCIS) residuals in breast
DFS | up to 2 years
  DFS defined as the time from drug onset until recurrence or death for various reasons.
Rate of breast conserving surgery | 3 months
  Rate of patients with breast conserving surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu J, He M, Ou K, Wang X, Wang Y, Qi L, Chai Y, Jiang M, Ma F, Luo Y, Yuan P, Zhang P, Xu B, Li Q. Efficacy and safety of apatinib combined with dose-dense paclitaxel and carboplatin in neoadjuvant therapy for locally advanced triple-negative breast cancer: A prospective cohort study with propensity-matched analysis. Int J Cancer. 2024 Jan 1;154(1):133-144. doi: 10.1002/ijc.34717. Epub 2023 Sep 7. PMID 37676110